CLINICAL TRIAL: NCT01792570
Title: Strategic Study of Dual-therapy With Darunavir/Ritonavir and Rilpivirine QD Versus Triple-therapy in Patients With Suppressed Viral Load: Virological Efficacy and Evaluation of Non-HIV Related Morbidity.
Brief Title: DRV/r + RPV QD: Efficacy and Toxicity Reduction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Collaborators: Elisa Colella, M.D. (Unknown); Valentina Di Cristo, M.D. (Unknown); Massimo Galli, M.D. (Unknown)
Responsible Party: Principal Investigator, Stefano Rusconi, Associate professor in infectious diseases, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HLS03/2012
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV-1; darunavir; rilpivirine; strategic study
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RPV + DRV/r (Experimental): switch to RPV + DRV/r
  Interventions: Drug: RPV + DRV/r
- continue the PI/r-containing HAART. (Active Comparator): continue the PI/r-containing HAART
  Interventions: Drug: continue the PI/r-containing HAART.

INTERVENTIONS:
Drug: RPV + DRV/r — Switch to dual HAART
  Other Names: RVP: rilpivirine; brand name: EdurantTM.; DRV: darunavir; brand name: PrezistaTM.
  Arms: RPV + DRV/r
Drug: continue the PI/r-containing HAART. — Continue the on-going triple drug HAART.
  Other Names: the drugs will depend on the successful regimen.
  Arms: continue the PI/r-containing HAART.

SUMMARY:
Clinical approach to HIV infection treatment is based on the use of highly active antiretroviral therapies (HAART) and recent national and international guidelines for guiding HIV therapy recommend the use of triple-combination therapy using antiretrovirals with 2 nucleos(t)ide inhibitors [N(n)RTI] as backbone plus a third drug to be chosen among a boosted protease inhibitor (PI/r), a nonnucleoside inhibitor (NNRTI) or an integrase inhibitor (II).

In spite of evident efficacy of HAART, as demonstrated by survival increasing, long term side effects, as for example the impact on renal function, remain principal problem.

In patient with risk factor for renal disease, a reduction of eGRF (estimated Glomerular Filtration Rate) between 90 and 60 mL/min/1,73 m2 could be already considered as a risk condition [1,2].

Efficacy of HAART, with increase of media survival and the parallel decrease of mortality, has underlined the necessity to reflect on long term HAART effects [3].

There are many evidences of HAART-related toxicity that, in spite of the necessity of a life-saving therapy, focus on the additional costs of this situation, in terms of health as well as in terms of economic costs.

Particular attention has been focused on the impact of some drugs on renal function, as tenofovir, especially on tubule, without forgetting the modification of lipid and bone metabolisms.

According to further studies which have evidenced the potential of some recently introduced molecules [4,5], the investigators had the need to realize a study to deepen the feasibility of a dual-therapy that permit to exclude NRTIs from the backbone, with the aim to prevent NRTIs-related long-term toxicity.

The investigators have designed a prospective randomized controlled trial, open-label, with a duration of 96 weeks, to compare the efficacy of a dual-therapy based on rilpivirine 25mg plus darunavir 800mg/ritonavir 100mg QD, in HIV-positive subjects with suppressed viremia from at least 3 months. In fact, there are a few data about association of these drugs, which it has been shown to be safe, well tolerated, and with a strong pharmacological synergy, without nucleos(t)idic backbone, while the necessity to minimize the costs toxicity-related is becoming increasingly compelling.

According to clinical experience and literature data, the investigators hope this study shows positive results in term of immune-virological efficacy, as well as in term of decrease of VACS index - a complex parameter which has the purpose to quantify general organic decay - and markers of lipid and bone metabolism, in group which receives dual-therapy versus the group with standard therapy.

DETAILED DESCRIPTION:
Pilot, phase III prospective, randomized, open-label, multicentric controlled study, which will offer a novel dual-therapy regimen including RPV 25mg + DRV 800mg/rtv 100mg QD to HIV+ subjects with suppressed viremia.

132 HIV+ subjects will be randomized, 1:1, to switch to RPV+DRV/r versus continue triple-drug therapy. Subjects will be switched from any PI/r-containing regimen.

The duration of the study is 96 weeks and patients will be stratified according to their HCV serostatus (Ab positive or negative), age (> or < 50 years), and immunological status (CD4<200/µL; CD4=200-500/µL; CD4>500/µL). It is planned to enroll at least 30% of female subjects.

Follow-up visits will be performed at 4, 8, 12, 24, 36, 48, 60, 72, and 96 weeks (laboratory and physical examination).

Effectiveness will be measured by determination of HIV-RNA, safety will be evaluated by determination of AST, ALT, creatinine, plasmatic and urinary phosphate, albuminuria, total cholesterol, HDL and LDL cholesterol, triglycerides at the follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult HIV+ subjects (>18 years old), giving and signing an informed consent;
* Any HAART treatment for at least 12 months;
* Current treatment with a PI/r-containing regimen initiated at least 6 months earlier;
* HIV-RNA <50 cp/mL for at least 3 months, without viral blip due to virologic failure at any time;
* Any nadir CD4 lymphocytes;
* Current CD4 count > 100 cell/uL;
* eGFRs >60 mL/min/1.73 m2.

Exclusion Criteria:

* Previous drug resistance genotypic test showing the presence of any RPV (RT: K101E/P, E138A/G/K/Q/R, V179L, Y181C/I/V, Y188L, H221Y, F227C, M230I/L) or DRV (protease: V11I, V32I, L33F, I47V, I50V, I54M/L, T74P, L76V, I84V, L89V) resistance associated mutation (RAM), according to the November 2011 IAS-USA list;
* Child-Pugh C or grade 3-4 AST or ALT values;
* Acute cardiovascular event within 6 months;
* AIDS event within 6 months;
* Current IVDU;
* HBsAg +;
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
HIV-RNA < 50 cp/mL | Week 48
  Responders: HIV+ subjects with HIV-RNA < 50 cp/mL at week 48 according to the intention-to-treat (ITT-TLOVR) approach.

SECONDARY OUTCOMES:
ACTG grade III and IV events. | over 96 weeks.
  Safety will be assessed through the number of ACTG grade III and IV in the specified safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Rusconi, M.D., Principal Investigator — DIBIC "Luigi Sacco", Università degli Studi di Milano, Italy
Locations (12):
- Italy (12):
  - Clinica delle Malattie Infettive, Policlinico Universitario, Bari, BA
  - Divisione di Malattie Infettive, Ospedale S. Maria Annunziata, Antella, Florence, FI
  - Clinica delle Malattie Infettive, Ospedale San Martino, Università degli Studi, Genova, GE
  - Divisione di Malattie Infettive, Ospedale San Gerardo, Monza, MB
  - Divisione Clinicizzata di Malattie Infettive dell'Università degli Studi, Dipartimento di Scienze Biomediche e Cliniche "Luigi Sacco", Milan, MI
  - I e II Divisione Malattie Infettive, Azienda Ospedaliera-Polo Universitario "Luigi Sacco", Milan, MI
  - Clinica Malattie Infettive, Policlinico Universitario, Modena, MO
  - U.O. Malattie Infettive, Policlinico S. Matteo, Pavia, PV
  - Clinica delle Malattie Infettive, Policlinico "Tor Vergata", Roma, RM
  - Istituto di Clinica delle Malattie Infettive, Università Cattolica del Sacro Cuore, Roma, RM
  - U.O. Malattie Infettive, Azienda Policlinico Umberto I, Università degli Studi "La Sapienza", Roma, RM
  - Clinica delle Malattie Infettive, Ospedale Amedeo di Savoia, Università degli Studi, Torino, TO

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Maggi P, Bartolozzi D, Bonfanti P, Calza L, Cherubini C, Di Biagio A, Marcotullio S, Montella F, Montinaro V, Mussini C, Narciso P, Rusconi S, Vescini F. Renal complications in HIV disease: between present and future. AIDS Rev. 2012 Jan-Mar;14(1):37-53. PMID 22297503
- [Background] Earley A, Miskulin D, Lamb EJ, Levey AS, Uhlig K. Estimating equations for glomerular filtration rate in the era of creatinine standardization: a systematic review. Ann Intern Med. 2012 Jun 5;156(11):785-95. doi: 10.7326/0003-4819-156-11-201203200-00391. Epub 2012 Feb 6. PMID 22312131
- [Background] Broder S. The development of antiretroviral therapy and its impact on the HIV-1/AIDS pandemic. Antiviral Res. 2010 Jan;85(1):1-18. doi: 10.1016/j.antiviral.2009.10.002. Epub 2009 Dec 16. PMID 20018391
- [Background] Burgos J, Crespo M, Falco V, Curran A, Imaz A, Domingo P, Podzamczer D, Mateo MG, Van den Eynde E, Villar S, Ribera E. Dual therapy based on a ritonavir-boosted protease inhibitor as a novel salvage strategy for HIV-1-infected patients on a failing antiretroviral regimen. J Antimicrob Chemother. 2012 Jun;67(6):1453-8. doi: 10.1093/jac/dks057. Epub 2012 Feb 29. PMID 22378681
- [Background] Clumeck N, Cahn P, Molina JM, Mills A, Nijs S, Vingerhoets J, Witek J. Virological response with fully active etravirine: pooled results from the DUET-1 and DUET-2 trials. Int J STD AIDS. 2010 Nov;21(11):738-40. doi: 10.1258/ijsa.2010.010139. PMID 21187353